CLINICAL TRIAL: NCT00466440
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase 2 Study With and Without Enzastaurin in Combination With Docetaxel and Prednisone, Followed By Enzastaurin Maintenance as First-Line Treatment in Hormone Refractory Metastatic Prostate Cancer Patients
Brief Title: A Phase 2 Study With Enzastaurin Plus Chemotherapy or Placebo Plus Chemotherapy for Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11311; H6Q-MC-S032 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzastaurin; Docetaxel; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- docetaxel + prednisone + enzastaurin (Experimental): Regimen A: docetaxel 75 milligrams per square meter (mg/m^2), intravenous (IV) is administered on Day 1 every 3 weeks for 6 cycles (maximum up to 10 cycles) and prednisone 5 milligrams (mg) oral (po), twice daily (BID) every day. In Cycle 1, enzastaurin is given as a loading dose of 1125 mg on the day prior to docetaxel and prednisone therapy, followed by enzastaurin 500 mg po, daily (QD) for the remaining Period 2 (chemotherapy) and Period 3 (maintenance).
  Interventions: Drug: enzastaurin; Drug: docetaxel; Drug: prednisone
- docetaxel + prednisone + placebo (Placebo Comparator): Regimen B: docetaxel 75 mg/m^2, IV is administered on Day 1 every 3 weeks for 6 cycles (maximum up to 10 cycles) and prednisone 5 mg po, BID every day. In Cycle 1, placebo is given as a loading dose on the day prior to docetaxel and prednisone therapy, followed by po, QD placebo for the remaining Period 2 (chemotherapy) and Period 3 (maintenance), until unblinding.
  Interventions: Drug: placebo
- docetaxel + prednisone + enzastaurin (modified Regimen A) (Experimental): Modified Regimen A, including pharmacokinetic (PK) characterization: Participants were treated with a modified investigational regimen with no dose escalation: docetaxel 75 mg/m2, IV was administered on Day 1 every 3 weeks for 6 cycles (maximum up to 10 cycles) and prednisone 5 mg po, BID every day. In Cycle 1, enzastaurin was given as a loading dose of 1125 mg starting on Day 4, followed by enzastaurin 500 mg po, QD for the remaining Period 2 (chemotherapy) and Period 3 (maintenance).
  Interventions: Drug: enzastaurin; Drug: docetaxel; Drug: prednisone

INTERVENTIONS:
Drug: enzastaurin — 1125 mg loading dose, then 500 mg po QD until disease progression, toxicity, or maximum 3 years
  Other Names: LY317615
  Arms: docetaxel + prednisone + enzastaurin; docetaxel + prednisone + enzastaurin (modified Regimen A)
Drug: placebo — Loading dose, then po QD until unblinding
  Arms: docetaxel + prednisone + placebo
Drug: docetaxel — 75 mg/m^2 IV, every 21 days, six 21-day cycles, maximum 10 cycles
  Arms: docetaxel + prednisone + enzastaurin; docetaxel + prednisone + enzastaurin (modified Regimen A)
Drug: prednisone — 5 mg po BID, six 21-day cycles
  Arms: docetaxel + prednisone + enzastaurin; docetaxel + prednisone + enzastaurin (modified Regimen A)

SUMMARY:
The purpose of the study is to compare the response rates for prostate cancer patients taking chemotherapy plus enzastaurin versus chemotherapy plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* You are at least 18 years old.
* You live close enough to the doctor's office to attend all of your required visits.
* You have not been treated with chemotherapy for your prostate cancer.
* Your organs must be functioning properly.

Exclusion Criteria:

* You are unable to swallow pills.
* You have another serious illness besides your prostate cancer.
* You have taken another experimental drug within the last 30 days.
* You have a serious heart condition.
* You are receiving another anti-cancer therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-06; Primary Completion 2009-08 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (28):
- United States (22):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fullerton, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northridge, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redondo Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Barbara, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Maria, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harvey, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Henderson, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Cruces, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport News, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Como
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Sisto

REFERENCES:
- [Derived] Dreicer R, Garcia J, Rini B, Vogelzang N, Srinivas S, Somer B, Shi P, Kania M, Raghavan D. A randomized, double-blind, placebo-controlled, Phase II study with and without enzastaurin in combination with docetaxel-based chemotherapy in patients with castration-resistant metastatic prostate cancer. Invest New Drugs. 2013 Aug;31(4):1044-50. doi: 10.1007/s10637-013-9940-0. Epub 2013 Feb 24. PMID 23435622
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Docetaxel + Prednisone + Enzastaurin: Participants were treated with modified Regimen A (modified investigational): docetaxel 75 milligrams per square meter (mg/m^2), intravenous (IV) given on Day 1 every 3 weeks, and prednisone 5 milligrams (mg) oral (po), twice daily (BID) in combination with enzastaurin, starting loading dose on Day 4.
- Part 2: Docetaxel + Prednisone + Enzastaurin: Regimen A: docetaxel 75 mg/m^2, IV given on Day 1 every 3 weeks and prednisone 5 mg po, BID with enzastaurin, starting loading dose 1 day prior to chemotherapy.
- Part 2: Docetaxel + Prednisone + Placebo: Regimen B: docetaxel 75 mg/m^2, IV is administered on Day 1 every 3 weeks for 6 cycles (maximum up to 10 cycles) and prednisone 5 mg po, BID every day. In Cycle 1, placebo is given as a loading dose on the day prior to docetaxel and prednisone therapy, followed by placebo po, QD for the remaining Period 2 (chemotherapy) and Period 3 (maintenance), until unblinding.
Period: Overall Study
Arm/Group | Part 1: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo
Started | 14 | 48 | 46
Received at Least One Dose of Study Drug | 14 | 47 | 41
Completed | 0 | 36 (Completed = completed 4 cycles of treatment) | 34 (Completed = completed 4 cycles of treatment)
Not Completed | 14 | 12 | 12
Not completed — Adverse Event | 0 | 3 | 1
Not completed — Death | 1 | 1 | 0
Not completed — Progressive disease | 13 | 5 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 2
Not completed — Protocol entry criteria not met | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Sponsor decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Docetaxel + Prednisone + Enzastaurin: Participants were treated with modified Regimen A (modified investigational): docetaxel 75 mg/m2 IV given on Day 1 every 3 weeks and prednisone 5 mg po BID in combination with enzastaurin, starting loading dose on Day 4.
- Part 2: Docetaxel + Prednisone + Enzastaurin: Regimen A: docetaxel 75 mg/m^2 IV given on Day 1 every 3 weeks and prednisone 5 mg po BID with enzastaurin, starting loading dose 1 day prior to chemotherapy.
- Part 2: Docetaxel + Prednisone + Placebo: Regimen B: docetaxel 75 mg/m^2 IV is administered on Day 1 every 3 weeks for 6 cycles (maximum up to 10 cycles) and prednisone 5 mg po BID every day. In Cycle 1, placebo is given as a loading dose on the day prior to docetaxel and prednisone therapy, followed by placebo po QD for the remaining Period 2 (chemotherapy) and Period 3 (maintenance), until unblinding.
- Total: Total of all reporting groups
Arm/Group | Part 1: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo | Total
Number analyzed (Participants) | 14 | 48 | 46 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (7.29) | 69.9 (7.66) | 70 (8.1) | 69.54 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 14 | 48 | 46 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 8 | 7 | 15
  White | 14 | 39 | 33 | 86
  Hispanic | 0 | 0 | 6 | 6
  East Asian | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 44 | 39 | 97
  Germany | 0 | 3 | 4 | 7
  Italy | 0 | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Percentage of Participants With Objective Tumor Response (Response Rate)
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST). Complete Response (CR)=disappearance of all target lesions; Partial Response (PR)=30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD)=20% increase in sum of longest diameter of target lesions; Stable Disease (SD)=small changes that do not meet above criteria. Objective response rate (%)=number of objective responders divided by the number of participants qualified for efficacy analysis *100, where objective responders are those participants who have met criteria either for CR or PR.
Time Frame: Baseline up to 3 years
Population: All enrolled participants from Part 2 group, who received at least one dose of study drug. Per protocol, Part 1 was not included as it is an open-label safety lead-in portion with PK characterization.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo
Number analyzed (Participants) | 46 | 40
percentage of participants | 15.2 [7.37 to 26.69] | 15.0 [6.74 to 27.47]
Statistical Analysis 1: Comparison: Part 2: Docetaxel + Prednisone + Enzastaurin vs Part 2: Docetaxel + Prednisone + Placebo; Test type: Superiority or Other; p = 1.0000, Chi-squared; Median Difference (Final Values) = 0.2, 90% CI 2-sided [-12.52 to 12.95] — The objective response rates and the 90% confidence intervals were estimated for the qualified participants using unadjusted normal approximation for binomial proportions (z approximation)

2. Secondary Outcome: Percentage of Participants Exhibiting a Decline in Prostate-Specific Androgen (PSA) From Baseline ≥30% Within First 3 Months of Treatment
Description: PSA is a protein produced by the cells of the prostate gland. PSA is present in small quantities in the serum of men with healthy prostates, but is often elevated in the presence of prostate cancer and in other prostate disorders. A blood test to measure PSA is considered the most effective test currently available for the early detection of prostate cancer. Decline in PSA of ≥30% from baseline within the first 3 months of treatment was calculated.
Time Frame: Baseline up to 3 months
Population: The analysis population included all participants having baseline and at least 1 postbaseline PSA response within the first 3 months of treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo
Number analyzed (Participants) | 9 | 28 | 29
percentage of participants | 69.2 [42.74 to 88.73] | 60.9 [47.68 to 72.97] | 72.5 [58.61 to 83.75]
Statistical Analysis 1: Comparison: Part 2: Docetaxel + Prednisone + Enzastaurin vs Part 2: Docetaxel + Prednisone + Placebo; Test type: Superiority or Other; p = 0.3606, Chi-squared; Mean Difference (Final Values) = -11.6, 90% CI 2-sided [-28.21 to 4.95]

3. Secondary Outcome: Prostate-Specific Androgen (PSA) Velocity at 2 Months
Description: PSA is a protein produced by the cells of the prostate gland. PSA is present in small quantities in the serum of men with healthy prostates, but is often elevated in the presence of prostate cancer and in other prostate disorders. A blood test to measure PSA is considered the most effective test currently available for the early detection of prostate cancer. PSA velocity is computed for each participant by means of linear regression on the logarithm of PSA. The linear regression fits a line through the logarithm of the PSA value on the y-axis, and the time from baseline on the x-axis with the baseline PSA value at time zero. The resulting slope is PSA velocity.
Time Frame: Baseline up to 2 months
Population: Participants with a valid baseline and at least 1 postbaseline PSA measurement within the first 2 months of treatment.
Measure: Mean (90% Confidence Interval); unit: microgram per liter (ug/L) per month
Arm/Group | Part 1: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo
Number analyzed (Participants) | 13 | 46 | 40
microgram per liter (ug/L) per month | -0.56 [-0.82 to -0.29] | -0.29 [-0.47 to -0.10] | -0.55 [-0.78 to -0.32]
Statistical Analysis 1: Comparison: Part 2: Docetaxel + Prednisone + Enzastaurin vs Part 2: Docetaxel + Prednisone + Placebo; Test type: Superiority or Other; p = 0.0720, t-test, 1 sided; Mean Difference (Final Values) = 0.26, 90% CI 2-sided [-0.02 to 0.55]

4. Secondary Outcome: Prostate-Specific Androgen (PSA) Velocity at 3 Months
Description: as for outcome 3
Time Frame: Baseline up to 3 months
Population: Participants with a valid baseline and at least 1 postbaseline PSA measurement within the first 3 months of treatment.
Measure: Mean (90% Confidence Interval); unit: ug/L per month
Arm/Group | Part 1: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo
Number analyzed (Participants) | 13 | 46 | 40
ug/L per month | -0.45 [-0.66 to -0.25] | -0.30 [-0.45 to -0.15] | -0.45 [-0.62 to -0.28]
Statistical Analysis 1: Comparison: Part 2: Docetaxel + Prednisone + Enzastaurin vs Part 2: Docetaxel + Prednisone + Placebo; Test type: Superiority or Other; p = 0.1697, t-test, 1 sided; Mean Difference (Final Values) = 0.15, 90% CI 2-sided [-0.07 to 0.37]

5. Secondary Outcome: Part 2: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of study enrollment to the first date of objectively determined progressive disease (PD) or death from any cause. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST version 1.0). PD is ≥20% increase in the sum of the longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. For participants not known to have died and who did not have PD, PFS was censored at the date of the last progression-free assessment. For participants who received subsequent systemic anticancer therapy (after discontinuation from the study treatment) prior to disease progression or death, PFS was censored at the date of last progression-free assessment prior to the initiation of post-discontinuation systemic anticancer therapy. No participant completed a full cycle of therapy and thus no formal analysis was performed.
Time Frame: Baseline to measured PD (up to 487 days)
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo
Number analyzed (Participants) | 46 | 40
Days | 229 [191 to 263] | 213 [188 to 240]
Statistical Analysis 1: Comparison: Part 2: Docetaxel + Prednisone + Enzastaurin vs Part 2: Docetaxel + Prednisone + Placebo; Test type: Superiority or Other; p = 0.5240, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.5 to 1.4]

6. Secondary Outcome: Part 2: Overall Survival (OS)
Description: Overall survival (OS) time is defined as the time from the date of diagnosis to the date of death from any cause. For participants who are still alive at the time of analysis, survival time will be censored at the last contact date.
Time Frame: Baseline to death (up to 642 days)
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo
Number analyzed (Participants) | 48 | 46
days | 462 [409 to 590] | 448 [383 to 453]
Statistical Analysis 1: Comparison: Part 2: Docetaxel + Prednisone + Enzastaurin vs Part 2: Docetaxel + Prednisone + Placebo; Test type: Superiority or Other; p = 0.4407, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.3 to 1.6]

7. Secondary Outcome: Part 2: Duration of Response
Description: Duration of response is defined as the time from date of objective response to progressive disease (PD) or death or prostate-specific androgen (PSA) returning to at least 50% from original baseline value.
Time Frame: First objective response to PD/death/PSA returning to 50% or more than the original baseline value (up to 616 days)
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo
Number analyzed (Participants) | 46 | 40
days | 231 [198 to 297] | 201 [175 to 225]
Statistical Analysis 1: Comparison: Part 2: Docetaxel + Prednisone + Enzastaurin vs Part 2: Docetaxel + Prednisone + Placebo; Test type: Superiority or Other; p = 0.3449, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.4 to 1.4]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A listing of serious AEs (SAEs) and all other non-serious AEs is included in the Reported Adverse Event Module.
Time Frame: Baseline through 3 years
Population: The analysis population was defined as all enrolled participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo
Number analyzed (Participants) | 14 | 47 | 41
Participants
  SAEs | 8 | 16 | 14
  Other Non-Serious AEs | 14 | 47 | 41

9. Secondary Outcome: Part I: Pharmacokinetic (PK) Parameter: Maximum Observed Drug Concentration During a Dosing Interval at Steady State (Cmax,ss) of Enzastaurin, LSN326020, and Total Analyte (Enzastaurin + LSN326020)
Description: Cmax,ss was calculated using concentration versus time data of enzastaurin, LSN326020, and total analyte (enzastaurin + LSN326020). Data are reported as Geometric Mean and Geometric Coefficient of Variation (%).
Time Frame: Part 1: Cycle 1, Day 21 - predose 2, 4, 6, 8, and 24 hours postdose; Cycle 2, Day 1 - predose, 2, 3, 4, 8, and 24 hours postdose
Population: For Part 1, pharmacokinetic analyses were conducted for individual participants who received at least one dose of study drug and had pharmacokinetic samples collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole per liter (nmol/L)
Groups:
- Enzastaurin 500 mg QD Alone: Enzastaurin, LSN326020 and total analyte (enzastaurin + LSN326020) on Cycle 1 Day 21 (enzastaurin alone) following enzastaurin 500 mg oral (po) daily (QD).
- Enzastaurin 500 mg QD + Docetaxel 75 mg/m^2 + Prednisone: Enzastaurin, LSN326020, and total analyte (enzastaurin + LSN326020) on Cycle 2 Day 1 (enzastaurin + docetaxel + prednisone) following enzastaurin 500 mg po QD.
Arm/Group | Enzastaurin 500 mg QD Alone | Enzastaurin 500 mg QD + Docetaxel 75 mg/m^2 + Prednisone
Number analyzed (Participants) | 9 | 7
nanomole per liter (nmol/L)
  Enzastaurin | 870 (84) | 778 (39)
  LSN326020 | 664 (45) | 667 (30)
  Total Analyte | 1540 (62) | 1450 (32)

10. Secondary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Concentration Versus Time Curve During 1 Dosing Interval at Steady State (AUCτ,ss) of Enzastaurin, LSN326020, and Total Analyte (Enzastaurin + LSN326020)
Description: AUCτ,ss was calculated using concentration versus time data of enzastaurin, LSN326020, and total analyte (enzastaurin + LSN326020). Data are reported as Geometric Mean and Geometric Coefficient of Variation (%).
Time Frame: Part 1: Cycle 1, Day 21 - predose 2, 4, 6, 8, and 24 hours postdose; Cycle 2, Day 1 - predose, 2, 3, 4, 8, and 24 hours postdose; Part 2: Cycle 2, Day 1 - predose, 1-3, and 4-9 hours postdose
Population: Pharmacokinetic analyses were conducted for individual participants who received at least one dose of study drug and had pharmacokinetic samples collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour per liter (nmol*hr/L)
Groups:
- Enzastaurin 500 mg QD Alone: Enzastaurin, LSN326020, and total analyte (enzastaurin + LSN326020) on Cycle 1 Day 21 (enzastaurin alone) following enzastaurin 500 mg oral (po) daily (QD).
- Enzastaurin 500 mg QD+Docetaxel 75 mg/m^2+Prednisone (Part 1); Enzastaurin 500 mg QD+Docetaxel 75 mg/m^2+Prednisone (Part 2): Enzastaurin, LSN326020, and total analyte (enzastaurin + LSN326020) on Cycle 2 Day 1 (enzastaurin + docetaxel + prednisone) following enzastaurin 500 mg po QD.
Arm/Group | Enzastaurin 500 mg QD Alone | Enzastaurin 500 mg QD+Docetaxel 75 mg/m^2+Prednisone (Part 1) | Enzastaurin 500 mg QD+Docetaxel 75 mg/m^2+Prednisone (Part 2)
Number analyzed (Participants) | 7 | 6 | 9
nanomole*hour per liter (nmol*hr/L)
  Enzastaurin | 12900 (79) | 13100 (26) | 20800 (104)
  LSN326020 | 15200 (35) | 15700 (20) | 24800 (52)
  Total Analyte | 28700 (49) | 29000 (18) | 47800 (74)

11. Secondary Outcome: Pharmacokinetic (PK) Parameter: Maximum Plasma Concentration (Cmax) of Docetaxel
Description: Cmax was calculated using concentration versus time data of docetaxel. Data are reported as Geometric Mean and Geometric Coefficient of Variation (%).
Time Frame: Part 1: Cycle 1, Day 1 - predose 0.5, 1, 1.5, 2, 3, 4, 8, and 24 hours postdose; Cycle 2, Day 1 - predose, 0.5, 1, 1.5, 2, 3, 4, 8, and 24 hours postdose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per millimeter (ng/mL)
Groups:
- Docetaxel 75 mg/m^2 Alone: Docetaxel (75 mg/m^2) following 1.0 hour intravenous infusion on Cycle 1 Day 1 (Docetaxel + Prednisone).
- Enzastaurin 500 mg QD + Docetaxel 75 mg/m^2 + Prednisone: Docetaxel (75 mg/m^2) following 1.0 hour intravenous infusion on Cycle 2 Day 1 (Docetaxel + Prednisone + Enzastaurin).
Arm/Group | Docetaxel 75 mg/m^2 Alone | Enzastaurin 500 mg QD + Docetaxel 75 mg/m^2 + Prednisone
Number analyzed (Participants) | 13 | 10
nanograms per millimeter (ng/mL) | 2230 (21) | 1840 (22)

12. Secondary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC[0-∞]) of Docetaxel
Description: AUC(0-∞) was calculated using concentration versus time data of docetaxel. Data are reported as Geometric Mean and Geometric Coefficient of Variation (%).
Time Frame: as for outcome 11
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Docetaxel 75 mg/m^2 Alone | Enzastaurin 500 mg QD + Docetaxel 75 mg/m^2 + Prednisone
Number analyzed (Participants) | 13 | 10
ng*h/mL | 2350 (26) | 1750 (20)

13. Secondary Outcome: Tumor Markers
Description: Pharmacogenomic (PGx) work on S032 was cancelled due to the limited number of tissue samples collected and the lack of clinical efficacy (responders) to enzastaurin. Potential biomarkers would have been assessed by dividing participants into low and high expression classes.
Time Frame: Baseline up to 36 months
Population: Data were not collected for any participant due to low samples.
Arm/Group | Part 1: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Part 1: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Enzastaurin | Part 2: Docetaxel + Prednisone + Placebo
Serious Adverse Events (participants affected / at risk) | 8/14 | 16/47 | 14/41
Other Adverse Events (participants affected / at risk) | 14/14 | 47/47 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Docetaxel + Prednisone + Enzastaurin (N=14) | Part 2: Docetaxel + Prednisone + Enzastaurin (N=47) | Part 2: Docetaxel + Prednisone + Placebo (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 6 (7) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Extravasation (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Docetaxel + Prednisone + Enzastaurin (N=14) | Part 2: Docetaxel + Prednisone + Enzastaurin (N=47) | Part 2: Docetaxel + Prednisone + Placebo (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 14 (17) | 7 (7)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 9 (35) | 5 (10)
Lymphopenia (Blood and lymphatic system disorders) | 9 (11) | 5 (7) | 11 (14)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 18 (55) | 14 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 4 (4) | 2 (4)
Cardio-Respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 3 (3) | 1 (1)
Strabismus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 3 (3) | 1 (1) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 8 (10) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 11 (16) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 22 (35) | 15 (20)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (5) | 4 (5)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 21 (33) | 11 (14)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 5 (5) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 14 (16) | 4 (4)
Asthenia (General disorders) | 0 (0) | 10 (13) | 3 (3)
Extravasation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (9) | 26 (34) | 25 (32)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 2 (2) | 3 (3)
Malaise (General disorders) | 0 (0) | 5 (6) | 2 (2)
Mucosal inflammation (General disorders) | 1 (1) | 2 (2) | 2 (2)
Oedema (General disorders) | 2 (2) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 8 (10) | 9 (10)
Pain (General disorders) | 1 (1) | 2 (2) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Opportunistic infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 6 (7) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 7 (10) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 9 (13) | 7 (8)
Blood albumin decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Blood calcium decreased (Investigations) | 3 (3) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 6 (7) | 6 (7) | 2 (2)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 3 (4) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (2) | 0 (0) | 1 (1)
Blood uric acid decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 1 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 5 (5) | 5 (5) | 9 (11)
Neutrophil count decreased (Investigations) | 3 (3) | 2 (6) | 4 (4)
Platelet count decreased (Investigations) | 1 (1) | 1 (2) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 4 (4) | 7 (7)
Weight increased (Investigations) | 0 (0) | 1 (1) | 3 (3)
White blood cell count decreased (Investigations) | 3 (4) | 4 (8) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 12 (16) | 15 (16)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 7 (9) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 14 (17) | 8 (13)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (6) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (8) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (7) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (9) | 8 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 3 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (8) | 7 (7)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 11 (16) | 9 (11)
Dysgeusia (Nervous system disorders) | 3 (3) | 14 (18) | 8 (8)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 6 (8) | 8 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (2) | 4 (4) | 2 (2)
Nocturia (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 4 (5)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (6) | 10 (11)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 9 (10) | 6 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12) | 21 (21) | 22 (23)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (11) | 10 (10)
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 5 (5)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 6 (8) | 3 (3)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 3 (4)
Thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days